CLINICAL TRIAL: NCT04964739
Title: Gender and Sex Hormone Influences on Cannabis Use Disorder Remission
Brief Title: Gender/Sex & CUD Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00110801; R01DA054617 (NIH)
Record Dates: First submitted 2021-07-11; First posted 2021-07-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use Disorder, Mild; Cannabis Use Disorder, Moderate; Cannabis Use Disorder, Severe
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy - Men (Other): 112 participants identifying as men will be enrolled in 8 weeks of behavioral treatment for cannabis use disorder (CUD). They will receive a motivational interviewing session with a therapist followed by 7 weekly online modules of CBT4CBT with continued monitoring and support from a therapist. Gender and hormonal factors will be examined as predictors of CUD remission and cannabis outcomes.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT4CBT)
- Cognitive Behavioral Therapy - Women (Other): 112 participants identifying as women will be enrolled in 8 weeks of behavioral treatment for CUD. They will receive a motivational interviewing session with a therapist followed by 7 weekly online modules of CBT4CBT with continued monitoring and support from a therapist. Gender and hormonal factors will be examined as predictors of CUD remission and cannabis outcomes.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT4CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT4CBT) — Participants will receive one therapist-led motivational interviewing/goal setting session followed by 7 sessions of computerized CBT4CBT.

SUMMARY:
Adults (ages 18+) who would like to reduce their cannabis use (N=224) will be enrolled in an 8-week treatment program. All participants will receive counseling (1 goals session with a therapist followed by 7 weekly computerized cognitive-behavioral therapy sessions). Detailed cannabis assessments (biological and self-report) will be conducted throughout treatment and at 1-, 2-, and 3-months post-treatment completion. Daily electronic diaries will be administered via text message to record detailed logs of cannabis use quantity and frequency. Salivary samples will be collected (and video observed) daily throughout treatment to analyze for progesterone.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in a research study (otherwise, will be referred to appropriate clinical services if seeking clinical care).
2. Meet current (within last 30 days) DSM-5 criteria for cannabis use disorder.
3. Submit a positive urine cannabinoid test during screening.
4. Interested in treatment for cannabis use disorder.

Exclusion Criteria:

1. Significant or acutely unstable medical or psychiatric problems (i.e., psychosis, mania) that would contraindicate research procedures, interfere with safety, compromise data integrity, or preclude consistent study participation.
2. The presence of any substance use disorder requiring a higher level of care.
3. Significant risk of homicide or suicide.
4. Pregnant, trying to become pregnant, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 224 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in remission | Week 4
  Remission is classified as the absence of DSM-5 cannabis use disorder symptoms (except cravings) as measured by semi-structured diagnostic interview.
Proportion of participants in remission | Week 8
  Remission is classified as the absence of DSM-5 cannabis use disorder symptoms (except cravings) as measured by semi-structured diagnostic interview.
Proportion of participants in remission | Week 12
  Remission is classified as the absence of DSM-5 cannabis use disorder symptoms (except cravings) as measured by semi-structured diagnostic interview.
Proportion of participants in remission | Week 16
  Remission is classified as the absence of DSM-5 cannabis use disorder symptoms (except cravings) as measured by semi-structured diagnostic interview.
Proportion of participants in remission | Week 20
  Remission is classified as the absence of DSM-5 cannabis use disorder symptoms (except cravings) as measured by semi-structured diagnostic interview.
Reduction in cannabis use days | 8 weeks of treatment
  Number of cannabis use days assessed via daily diaries during treatment
Reduction in cannabis use episodes | 8 weeks of treatment
  Number of cannabis use episodes assessed via daily diaries during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Tomko, PhD, Principal Investigator — Medical University of South Carolina; Aimee L McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators support data sharing as essential for scientific advancement. It is expected that primary outcome papers will be completed and submitted to appropriate peer-reviewed scientific journals within 180 days of data lock. Requests for data from this project by individuals outside of the research team will be reviewed by the team following data lock. Data sharing will adhere to all provisions of the Health Insurance Portability and Accountability Act (HIPAA) and the rights and privacy of people who participate in research will be protected at all times. The requesting Investigator must specify the subset of variables needed or provide a detailed justification of why the complete dataset is absolutely necessary. Data made available to other investigators will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects.

DOCUMENTS (1):
  • Informed Consent Form (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04964739/ICF_001.pdf